CLINICAL TRIAL: NCT04023110
Title: A Pilot Study of Risk-Guided Cardioprotection With Carvedilol in Breast Cancer Patients Treated With Doxorubicin and/or Trastuzumab
Brief Title: Risk-Guided Cardioprotection With Carvedilol in Breast Cancer Patients Treated With Doxorubicin and/or Trastuzumab
Acronym: CCTGuide Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPCC12118; R21HL150723 (NIH); 849569 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2019-03-22; First posted 2019-07-17 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Cardiotoxicity; Risk Factor, Cardiovascular; Toxicity Due to Chemotherapy; Breast Cancer; Cardiomyopathies; Heart Failure
Keywords: Risk-Guided Intervention; Carvedilol; Cardiotoxicity of Chemotherapy; Cardio-Oncology; Cardiomyopathy
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms; Cardiomyopathies; Heart Failure | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: An internally validated CV risk score will be used to determine an individual patient's risk. Low risk patients will be observed and managed according to usual care. Elevated risk patients will be randomized to open label, individually dosed carvedilol for 1 year or usual care.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol will be initiated at 3.125mg twice daily and uptitrated as tolerated in a stepwise fashion to a maximum dose of 25mg twice daily or to a systolic blood pressure (SBP) of 110-120mmHg or heart rate (HR) of 50-55 beats per minute (bpm). Patients will start carvedilol in the evening after first dose of chemotherapy and will continue on medication for 12 months.
  Clinical, echocardiographic, and biomarker data will be collected on all patients at baseline and standardized time intervals during and after therapy at approximately 3, 6, 9, 12, and 24 months.
  Interventions: Drug: Carvedilol
- Usual Care (No Intervention): Clinical, echocardiographic, and biomarker data will be collected on all patients at baseline and standardized time intervals during and after therapy at approximately 3, 6, 9, 12, and 24 months.

INTERVENTIONS:
Drug: Carvedilol — Individually dosed carvedilol
  Other Names: Coreg
  Arms: Carvedilol

SUMMARY:
Investigators will evaluate the safety, tolerability, and feasibility of a risk-guided cardioprotective treatment strategy with carvedilol, as compared to usual care, in breast cancer patients undergoing treatment with doxorubicin, trastuzumab, or the combination.

DETAILED DESCRIPTION:
This is a single-center, randomized clinical trial that seeks to determine if a risk guided treatment strategy that initiates carvedilol in high risk breast cancer patients prior to doxorubicin and/or trastuzumab is safe, tolerable, and feasible. Subjects who are identified as having elevated CTX Risk by an internally validated clinical risk score (exceeding a pre-specified risk threshold) will be randomized to individually-dosed, open-label carvedilol or usual care. Investigators will use a stratified randomization according to trastuzumab therapy (yes/no) to ensure balance across treatment regimen. Clinical, echocardiographic, and biomarker data will be collected on all patients at baseline and standardized time intervals during and after therapy at approximately 3, 6, 9, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Females
* At least 18 years old
* Diagnosed with Stage I-III breast cancer with treatment plan to include therapy with anthracyclines and/or trastuzumab in the adjuvant or neo-adjuvant setting
* Study team is able to obtain all necessary information for calculating Cardiotoxicity Risk Score (including echocardiographic measurement of left ventricular ejection fraction)

Exclusion Criteria:

* Pregnant or breast feeding. Due to unknown risks and potential harm to the unborn fetus a negative pregnancy test within 10 days prior to enrollment is required in women with child-bearing potential. Due to the potential nursing infant harm, women who are currently breast feeding are not eligible for this study.
* Contraindication to carvedilol
* Baseline systolic blood pressure < 90mmHg (if multiple blood pressures are available in the medical record within 1 month prior to screening, the average SBP will be considered)
* Baseline heart rate < 55 bpm consistent with severe bradycardia (if multiple resting heart rates are available in the medical record within 1 month prior to screening, the average heart rate will be considered)
* Allergy to carvedilol
* History of bronchial asthma or related bronchospastic conditions
* Known history of sick sinus syndrome
* Severe hepatic impairment, defined as serum bilirubin > 3.0x ULN, AST or ALT > 5.0 ULN within 28 days of enrollment
* Second- or third-degree AV block, as determined by electrocardiogram
* Severe bradycardia (unless permanent pacemaker is in place)
* Patients in cardiogenic shock or decompensated heart failure requiring the use of IV inotropic therapy
* Current use of: Bupropion (Wellbutrin), Fluoxetine (Prozac), Paroxetine (Paxil), Quinidine (Quinidex), Duloxetine (Cymbalta), Digoxin
* Current treatment with beta blocker
* Unable to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, MSCE, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to make the IPD, analytic methods, or study materials available to other researchers for purposes of reproducing our results or replicating the procedure given the pilot Phase 1 nature of this study.

REFERENCES:
- [Derived] Jung W, Hubbard RA, Smith AM, Ko K, Huang A, Wang J, Isaacs JM, Zhang L, Liu PP, Chen Z, Shah PD, Mintzer D, Bhattacharya S, Knollman HM, Clark AS, Koropeckyj-Cox D, Messinger M, Wilcox NS, Xia C, Narayan V, Upshaw JN, Armenian SH, Ky B. Risk-guided cardioprotection with carvedilol in patients with breast cancer (CCT guide): a phase 1 randomized clinical trial. Breast Cancer Res Treat. 2025 Jun;211(2):293-305. doi: 10.1007/s10549-025-07636-3. Epub 2025 Apr 2. PMID 40172740

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The cardiotoxicity risk score was calculated using Cox proportional hazards regression with race, systolic blood pressure, left ventricular ejection fraction, systemic cancer therapy, smoking status, diabetes and hypertension as selected predictors (PMID 4012740). A threshold of 4.5% risk of cardiac dysfunction at 1 year was set to prioritize sensitivity. 49 patients were classified as low risk and 19 as elevated risk. 13 elevated risk patients were randomized to carvedilol and 6 to usual care.
Groups:
- Elevated Risk / Carvedilol: Patients determined to be elevated risk and randomized to carvedilol (elevated risk/carvedilol arm) initiated carvedilol at a dose of 3.125 mg twice daily on the evening of the first cancer therapy cycle and continued for 12 months. Dose adjustments were based on tolerability and targeted parameters as determined by the study physician, and carvedilol was titrated to maximum tolerated dose by the participant or to a SBP of 110-120mmHg or heart rate (HR) of 50-55 beats per minute. Titration steps were predefined at doses of 6.25 mg, 12.5 mg, and up to 25 mg twice daily. Clinical, echocardiographic, and biomarker data were collected at baseline and standardized time intervals during and after therapy at approximately 3, 6, 9 12 and 24 months.
- Elevated Risk/Usual Care: Patients with elevated risk who were randomized to the Elevated Risk/Usual Care arm were followed with clinical, echocardiographic, and biomarker data collected at baseline and standardized time intervals during and after therapy at approximately 3, 6, 9, 12, and 24 months.
- Low Risk / Non-randomized: Patients who did not meet the threshold for elevated risk were not randomized, but were followed with clinical, echocardiographic, and biomarker data collected at baseline and standardized time intervals during and after therapy at approximately 3, 6, 9, 12, and 24 months.
Period: Overall Study
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Started | 13 | 6 | 49
12 Month | 10 | 6 | 47
24 Month | 10 | 6 | 47
Completed | 10 | 6 | 47
Not Completed | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized | Total
Number analyzed (Participants) | 13 | 6 | 49 | 68
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [47 to 62] | 51 [47 to 56] | 52 [41 to 60] | 52 [42 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 49 | 68
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Race and ethnicity were self-reported
  Participants
    Hispanic or Latino | 0 | 1 | 0 | 1
    Not Hispanic or Latino | 13 | 5 | 49 | 67
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race and ethnicity were self-reported.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 4 | 17 | 24
    White | 7 | 1 | 29 | 37
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 2 | 1 | 2 | 5
Systolic Blood Pressure (SBP) [Median (Inter-Quartile Range); unit: mmHg] | 127 [105 to 149] | 121 [114 to 138] | 125 [117 to 136] | 125 [116 to 138]
Left Ventricular Ejection Fraction (LVEF) [Median (Inter-Quartile Range); unit: percent] — LVEF by echocardiogram. Left ventricular ejection fraction (LVEF) is defined as the left ventricular stroke volume (left ventricular end diastolic volume minus the left ventricular end systolic volume) divided by the left ventricular end diastolic volume. This fraction is multiplied by 100 to yield the LVEF, and is defined as a % (the unit of measure) (J Am Soc Echocardiogr 2015;28:1-39.). 2D left ventricular volumes are estimated according to the biplane method of disks (modified Simpson's rule), as recommended by societal guidelines. Higher values are generally considered more favorable.
  percent | 61.1 [58.2 to 64.8] | 59.6 [57.6 to 59.9] | 61.9 [60.0 to 65.0] | 61.2 [59.3 to 64.8]
Systemic Cancer Therapy (Anthracyclines and Her2 targeted agents) [Count of Participants; unit: Participants] — Patient received a systemic therapy regimen containing doxorubicin or Her2 targeted therapy or the combination.
  Participants
    Doxorubicin | 10 | 4 | 26 | 40
    Her2 Targeted | 2 | 1 | 23 | 26
    Doxorubicin + Her2 Targeted | 1 | 1 | 0 | 2
Smoking Status [Count of Participants; unit: Participants] — Current and prior smokers
  Participants | 6 | 2 | 14 | 22
Diabetes [Count of Participants; unit: Participants] | 2 | 1 | 2 | 5
Hypertension (HTN) [Count of Participants; unit: Participants] — Patients were considered to have HTN at baseline if they had a diagnosis of hypertension, or were taking anti-hypertensives, or had systolic blood pressure > 140 on average over the 6 weeks prior to enrollment.
  Participants | 2 | 2 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF by echocardiogram. Left ventricular ejection fraction (LVEF) is defined as the left ventricular stroke volume (left ventricular end diastolic volume minus the left ventricular end systolic volume) divided by the left ventricular end diastolic volume. This fraction is multiplied by 100 to yield the LVEF, and is defined as a % (the unit of measure) (J Am Soc Echocardiogr 2015;28:1-39.). 2D left ventricular volumes are estimated according to the biplane method of disks (modified Simpson's rule), as recommended by societal guidelines. Higher values are generally considered more favorable.
Time Frame: up to 24 months
Population: Exploratory cardiac efficacy by cardiac function (LVEF) was analyzed, evaluating the three groups according to the treatment the participants actually received ("as treated").
  After randomization, three participants refused carvedilol but agreed to remain on study for follow-up, and one participant assigned to usual care started carvedilol for clinical indications at the baseline visit. As a result, there were 11 participants treated with carvedilol and 8 treated as per usual care.
Measure: Median (Inter-Quartile Range); unit: percent
Groups:
- Elevated Risk / Carvedilol: Carvedilol will be initiated at 3.125mg twice daily and uptitrated as tolerated in a stepwise fashion to a maximum dose of 25mg twice daily or to a systolic blood pressure (SBP) of 110-120mmHg or heart rate (HR) of 50-55 beats per minute (bpm). Patients will start carvedilol in the evening after first dose of chemotherapy and will continue on medication for 12 months.
  Clinical, echocardiographic, and biomarker data will be collected on all patients at baseline and standardized time intervals during and after therapy at approximately 3, 6, 9, 12, and 24 months.
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
percent
  Baseline | 61.1 [59.7 to 64.9] | 59.0 [57.2 to 60.4] | 61.9 [60.0 to 65.0]
  12 Month | 58.4 [57.4 to 59.3] | 60.4 [59.1 to 61.9] | 59.7 [56.9 to 62.3]
  24 Month | 61.7 [57.3 to 62.3] | 61.7 [59.4 to 62.5] | 60.3 [58 to 62.6]

2. Primary Outcome: Treatment Adherence as Measured by Pill Count
Description: Rate of compliance with prescribed dose of carvedilol assessed based on pill count. Patients in the elevated-risk carvedilol group were asked to bring their study medications to all study visits and remaining pills were counted by the study coordinator to determine how many pills had been taken. Treatment adherence was calculated as the ratio of number of pills taken to expected number of pills taken, and is reported as a percentage. An adherence rate closer to 100 is better.
  Treatment adherence is reported only for those patients who were assigned to the elevated risk/carvedilol group, and therefore expected to take study medication.
Time Frame: 12 months
Population: Adherence to the carvedilol intervention was calculated only among the elevated-risk carvedilol group.
Measure: Median (Full Range); unit: percent of prescribed doses
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 13 | 0 | 0
percent of prescribed doses | 93 [0 to 99.4] |  |

3. Primary Outcome: Adverse Events
Description: Targeted Adverse Events were prospectively assessed according to the CTCAE v5.0. The number of patients experiencing any adverse event (Grade 2-5) was tabulated by risk group and by treatment arm during carvedilol intervention (baseline - 12 months). In the CTCAE, grade refers to the severity of the event. Grade 2 events are moderate, or have non-urgent/non-invasive intervention indicated, or limit age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 events are severe/medically significant but not immediately life-threatening, or have hospitalization or prolongation of hospitalization indicated, or limit self-care ADLs. Grade 4 events have life-threatening consequences or have urgent intervention indicated. Grade 5 indicates a death related to the adverse event.
Time Frame: Up to 12 months
Population: Safety was analyzed, evaluating the three groups according to the treatment the participants actually received ("as treated").
  After randomization, three participants refused carvedilol but agreed to remain on study for follow-up, and one participant assigned to usual care started carvedilol for clinical indications at the baseline visit. As a result, there were 11 participants treated with carvedilol and 8 treated as per usual care.
Measure: Count of Participants; unit: Participants
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
Participants
  Grade 2 and Higher | 11 | 8 | 47
  Grade 3 and Higher | 6 | 2 | 15
  Grade 4 and Higher | 1 | 0 | 1
  Grade 5 | 1 | 0 | 1

4. Secondary Outcome: Diastolic Function (E/e') by Echocardiogram
Description: E/e' is a measure of diastolic function derived from the ratio of the pulse wave Doppler interrogations of the mitral inflow at the mitral valve leaflet tips and at the lateral and septal mitral annulus via tissue Doppler imaging. This measure provided insight into myocardial relaxation, preload, and left ventricular filling pressures, with values > 14 indicative of elevated filling pressure. This is core-lab quantified, blinded to patient and treatment characteristics.
Time Frame: up to 24 months
Population: Exploratory cardiac efficacy by diastolic function was analyzed, evaluating the three groups according to the treatment the participants actually received ("as treated").
  After randomization, three participants refused carvedilol but agreed to remain on study for follow-up, and one participant assigned to usual care started carvedilol for clinical indications at the baseline visit. As a result, there were 11 participants treated with carvedilol and 8 treated as per usual care.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
ratio
  Baseline | 7.86 [6.89 to 8.60] | 6.85 [6.07 to 7.78] | 7.64 [6.54 to 8.70]
  12 Month | 8.22 [7.65 to 9.18] | 8.24 [6.79 to 8.82] | 7.06 [6.46 to 8.45]
  24 Month | 8.25 [7.05 to 8.67] | 7.90 [7.20 to 8.68] | 7.04 [6.43 to 7.99]

5. Secondary Outcome: Ventricular-arterial Coupling Measured by Echocardiogram
Description: Ventricular-arterial (VA) coupling, the ratio between effective arterial elastance (Ea), indicative of load, and end-systolic elastance (Ees), indicative of LV contractility, was also quantified. Ea/Ees is a measure of cardiac efficiency, with normal values of 0.8-1.0, and lower numbers typically indicative of greater efficiency and higher values reflective of worse function. This is core-lab quantified, blinded to patient and treatment characteristics.
Time Frame: up to 24 months
Population: Exploratory cardiac efficacy by ventricular arterial coupling was analyzed, evaluating the three groups according to the treatment the participants actually received ("as treated").
  After randomization, three participants refused carvedilol but agreed to remain on study for follow-up, and one participant assigned to usual care started carvedilol for clinical indications at the baseline visit. As a result, there were 11 participants treated with carvedilol and 8 treated as per usual care.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
ratio
  Baseline | 0.76 [0.62 to 0.83] | 0.84 [0.68 to 0.95] | 0.71 [0.58 to 0.92]
  12 Month | 0.83 [0.64 to 0.94] | 0.88 [0.84 to 0.89] | 0.82 [0.71 to 0.93]
  24 Month | 0.83 [0.78 to 0.94] | 0.78 [0.74 to 0.89] | 0.82 [0.71 to 0.96]

6. Secondary Outcome: Cardiac Strain Measurements by Echocardiogram
Description: Global longitudinal strain (GLS, %) averaged from 3 apical views (left ventricular apical 4-chamber, 2-chamber, and 3-chamber) was obtained using speckle-tracking technology using Tomtec Imaging Systems. GLS is a more sensitive measure of cardiac function, with values greater than -16% (e.g., -15%) for GLS associated with worse outcomes.
  Circumferential strain (GCS, %) from the short axis view (mid left ventricle) was obtained using speckle-tracking technology using Tomtec Imaging Systems. Circumferential strain is a more sensitive measure of cardiac function, with values or greater than -20% (e.g., -19%) associated with worse outcomes.
  GLS and GCS are core-lab quantified, blinded to patient and treatment characteristics.
Time Frame: up to 24 months
Population: Exploratory cardiac efficacy by longitudinal strain was analyzed, evaluating the three groups according to the treatment the participants actually received ("as treated").
  After randomization, three participants refused carvedilol but agreed to remain on study for follow-up, and one participant assigned to usual care started carvedilol for clinical indications at the baseline visit. As a result, there were 11 participants treated with carvedilol and 8 treated as per usual care.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
percent
  Baseline GLS | -20.7 [-21.8 to -20.2] | -20.5 [-23.0 to -20.1] | -21.8 [-22.9 to -20.6]
  12 Month GLS | -21.1 [-22.6 to -20.0] | -20.0 [-21.6 to -19.4] | -21.3 [-23.2 to -19.8]
  24 Month GLS | -22.0 [-22.9 to -20.3] | -22.1 [-25.3 to -20.2] | -21.3 [-22.6 to -20.0]
  Baseline GCS | -29.0 [-34.4 to -24.3] | -24.4 [-27.5 to -22.7] | -27.9 [-30.6 to -23.4]
  12 Month GCS | -24.3 [-25.3 to -22.9] | -26.2 [-30.1 to -23.6] | -25.2 [-28.2 to -21.9]
  24 Month GCS | -25.0 [-27.9 to -22.5] | -24.7 [-29.7 to -22.3] | -27.2 [-31.1 to -23.3]

7. Secondary Outcome: Frequency of Individuals With Cardiac Dysfunction
Description: Frequency of individuals with cardiac dysfunction, as defined by reduction in LVEF of >/= 10% to < 50%.
Time Frame: up to 24 months
Population: Exploratory cardiac efficacy was analyzed, evaluating the three groups according to the treatment the participants actually received ("as treated").
  After randomization, three participants refused carvedilol but agreed to remain on study for follow-up, and one participant assigned to usual care started carvedilol for clinical indications at the baseline visit. As a result, there were 11 participants treated with carvedilol and 8 treated as per usual care.
Measure: Count of Participants; unit: Participants
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
Participants | 0 | 0 | 1

8. Secondary Outcome: High-sensitivity Troponin (hsTnT) Level
Description: Change in the cardiac biomarker of injury hsTnT over time, defined as a continuous variable. hsTnT is a biomarker that is indicative of cardiac injury, with higher values associated with more severe injury. This is core-lab quantified, blinded to patient and treatment characteristics.
Time Frame: up to 24 months
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
ng/L
  Baseline | 6.1 [4.7 to 7.3] | 8.0 [6.4 to 8.4] | 5.7 [4.1 to 8.0]
  12 Month | 7.4 [6.4 to 8.0] | 6.2 [4.2 to 8.7] | 7.2 [5.6 to 9.4]
  24 Month | 7.0 [5.6 to 8.0] | 6.0 [4.7 to 7.3] | 6.4 [5.3 to 8.2]

9. Secondary Outcome: N-terminal Pro B-type Natriuetic Peptide (NTproBNP) Level
Description: Change in the cardiac biomarker, NT-proBNP over time, defined as a continuous variable. NTproBNP is a biomarker that is indicative of neurohormonal stress, with higher levels associated with more neurohormonal stress. This is core-lab quantified, blinded to patient and treatment characteristics.
Time Frame: up to 24 months
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
ng/L
  Baseline | 88.4 [57.1 to 100.1] | 54.8 [43.2 to 74.3] | 98.4 [35.5 to 161.6]
  12 Month | 126.8 [23.2 to 143.9] | 32.6 [19.6 to 82.7] | 52.0 [25.3 to 108.9]
  24 Month | 81.7 [54.9 to 110.5] | 53.9 [33.6 to 91.6] | 46.6 [30.1 to 113.5]

10. Secondary Outcome: Left Ventricular Mass
Description: LV mass by echocardiogram. Measurements of left ventricular mass (g) provided insight into cardiac structure, size, and remodeling. LV mass was calculated by the area-length method, as recommended by societal guidelines. This is core-lab quantified, blinded to patient and treatment characteristics.
Time Frame: up to 24 Months
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
Number analyzed (Participants) | 11 | 8 | 49
g
  Baseline | 110.6 [87 to 124.9] | 95.3 [87.2 to 103.6] | 98 [84.5 to 120]
  12 Month | 92.2 [75.4 to 103.6] | 98.4 [90.2 to 138.0] | 94.5 [84.2 to 112.2]
  24 Month | 80.2 [65.6 to 91.9] | 96.9 [85.8 to 120.8] | 97.8 [90 to 108.5]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse Events were assessed and graded according to the CTCAE v5.0. At each visit, patients were assessed for grade 2 and higher targeted adverse events (bradycardia, fatigue, and hypotension) as well as cardiovascular events and events ending in death using chart review and patient interview. All SAEs and AEs collected as part of the study and consistent with reporting requirements are reported.
Arm/Group | Elevated Risk / Carvedilol | Elevated Risk/Usual Care | Low Risk / Non-randomized
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/8 | 1/49
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/8 | 1/49
Other Adverse Events (participants affected / at risk) | 11/11 | 8/8 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elevated Risk / Carvedilol (N=11) | Elevated Risk/Usual Care (N=8) | Low Risk / Non-randomized (N=49)
Disease Progression (General disorders) | 1 | 0 | 0 — unrelated to intervention
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 — Unrelated to intervention (COVID-19 related)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elevated Risk / Carvedilol (N=11) | Elevated Risk/Usual Care (N=8) | Low Risk / Non-randomized (N=49)
Hypertension (Vascular disorders) | 9 | 3 | 30 — Grade 2 and higher
Fatigue (General disorders) | 4 | 4 | 23 — Grade 2 and higher
Ejection Fraction Decreased (Investigations) | 0 | 0 | 8 — Grade 2 and higher
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 0 | 8 — Grade 2 and higher
Thromboembolic Event (Vascular disorders) | 0 | 1 | 6 — Grade 2 and higher
Dizziness (Nervous system disorders) | 0 | 0 | 4 — Grade 2 and higher
Hypotension (Vascular disorders) | 0 | 0 | 3 — Grade 2 and higher
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 3 — Grade 2 and higher
Pre-Syncope (Nervous system disorders) | 1 | 1 | 1 — Grade 2 and higher

LIMITATIONS AND CAVEATS:
The limitations include small sample size and the fact that concomitant use of cardiac medications was not controlled. The study was executed during the COVID-19 pandemic which may have impacted patient recruitment and adherence.

Hypothesis testing was not conducted due to the limited sample size and exploratory nature of the study. Descriptive summary statistics were used to characterize the study population, outcome measures, and adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT04023110/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT04023110/ICF_001.pdf